CLINICAL TRIAL: NCT01391611
Title: A Phase II Study of Pazopanib in Patients With Imatinib Refractory or Intolerant Gastrointestinal Stromal Tumors (GIST)
Brief Title: Pazopanib in Imatinib Refractory or Intolerant Gastrointestinal Stromal Tumors (GIST)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy - Futility endpoint reached
Sponsor: Kristen Ganjoo (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Kristen Ganjoo, Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20636; RR2002/00017/09 (Other: GlaxoSmithKline); 11-311 (Other: Stanford IRB alternate); GIST0003 (Other: OnCore)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2016-12

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib arm (Experimental)
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 800 mg; PO
  Other Names: Votrient

SUMMARY:
This study is being done to gather information about the safety (any harmful effects) and effectiveness (usefulness) of Pazopanib in the treatment of Gastrointestinal Stroma Tumors (GIST) that cannot be treated by surgery or has spread to other organs. The Food and Drug Administration (FDA) have approved Pazopanib for the treatment of advanced kidney cancer but it is not approved for the treatment of GIST. The investigators hope to learn about the safety and usefulness (effectiveness) of Pazopanib for patients with GIST.

Primary Objective:

Non-progression rate based on RECIST criteria (CR+PR+SD)

Secondary Objectives:

* Response per Choi criteria
* 6 month progression-free survival
* Safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable gastrointestinal stromal tumor (GIST)
* Failure or intolerance to Imatinib and sunitinib
* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up.
* Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Measurable disease criteria by RECIST criteria
* Adequate organ system function as defined in protocol.
* A female is eligible to enter and participate in this study if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant). This includes any female who has had:
* A hysterectomy
* A bilateral oophorectomy (ovariectomy)
* A bilateral tubal ligation
* Menopause
* Childbearing potential females must have a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agree to use adequate contraception. Adequate acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
* An intrauterine device with a documented failure rate of less than 1% per year.
* Vasectomized partner who is sterile prior to the female subject?s entry and is the sole sexual partner for that female.
* Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.

Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide edify eligible disease(s)/stage(s)

Exclusion Criteria:

* History of other malignancies within 5 years prior to Day 1 except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma, squamous-cell carcinoma of the skin, carcinoma in situ of the cervix, early-stage bladder cancer, or low-grade endometrial cancer
* Clinically significant gastrointestinal abnormalities that may affect absorption of the investigational product
* Presence of uncontrolled infection
* Prolongation of corrected QT interval (QTc) > 480 milliseconds. On antiarrhythmics or medications known to prolong QT interval
* History of any one or more of the following cardiovascular conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Coronary artery by-pass graft surgery
* Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of >=140 mmHg or diastolic blood pressure (DBP) of >= 90mmHg].
* History of cerebrovascular accident, hemoptysis, cerebral hemorrhage, clinically significant GI bleed, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture
* Evidence of active bleeding or bleeding diathesis.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to procedures.
* Patients on strong CYP3A4 inhibitors
* Uncorrected abnormal electrolytes- K, Mg and Ca
* Treatment with any of the following anti-cancer therapies:
* o radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
* o chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen N. Ganjoo, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pazopanib Arm
Started | 25
Completed | 3
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib Arm
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 59 [27 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 18
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Non-progression Rate Based on RECIST 1.0 Criteria (CR+PR+SD)
Description: 4-mo non-progression rate
  "Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: 24 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib Arm
Number analyzed (Participants) | 25
months | 1.9 [1.6 to 5.2]

2. Secondary Outcome: Response Per Choi Criteria
Description: Response per Choi criteria
  * Complete response - Disappearance of all lesions; no new lesion
  * Partial response - A decrease in size of > or = 10% or a decrease in tumor density (HU) > or = 15% on CT. No new lesions. No obvious progression of nonmeasurable disease.
  * Stable disease - Does not meet the criteria for CR, PR, or PD. No symptomatic deterioration attributed to tumor progression.
  * Progressive disease - An increase in tumor size of > or = 10% and does not meet criteria of PR by tumor density (HU) on CT. New lesions. New intratumoral nodules or increase in the size of the existing intratumoral nodules.
Time Frame: 6 months
Population: Choi criteria measurements were not done due to technical difficulties.
Arm/Group | Pazopanib Arm
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Time Frame: All adverse events (related and unrelated) occurring during the study (from the time the patient receives the first dose of study drug) and up to 30 days after the last dose of study medication were reported. These were captured every months at clinic visit and patients also could report in between visits.
Description: Patients were asked about adverse events at every clinic visit.
Arm/Group | Pazopanib Arm
Serious Adverse Events (participants affected / at risk) | 14/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib Arm (N=25)
Worsened shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism G3 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Worsened ascites G1 (Gastrointestinal disorders) | 1 (1)
Deep venous thrombosis G1 (Vascular disorders) | 1 (1)
Pneumonia G1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Worsened right pleural effusion G1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
General disorders and administration site conditions-other, specify, Disease progression-fatal G5 (General disorders) | 1 (1)
Constipation G2 (Gastrointestinal disorders) | 1 (1)
GI disorders-other, E. coli bacteremia G3 (Gastrointestinal disorders) | 1 (1)
Intestinal perforation G4 (Gastrointestinal disorders) | 1 (1)
Fatigue G2 (General disorders) | 1 (1)
Sacral decubitus G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Ascites G3 (Gastrointestinal disorders) | 2 (2)
Peripheral motor neuropathy G2 (Nervous system disorders) | 1 (1)
Seizure G3 (Nervous system disorders) | 1 (1)
Nonviral hepatitis/transaminitis G2 (Hepatobiliary disorders) | 1 (1)
Anemia G2 (Blood and lymphatic system disorders) | 1 (1)
Hypoalbuminemia G3 (Metabolism and nutrition disorders) | 1 (1)
Worsening fatigue G3 (General disorders) | 1 (1)
Abdominal pain G3 (Gastrointestinal disorders) | 2 (4)
Dehydration G3 (Metabolism and nutrition disorders) | 1 (1)
Renal failure G5 (Renal and urinary disorders) | 1 (1)
GI Bleed G3 (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage, rectum bleeding (Gastrointestinal disorders) | 1 (1)
GI Bleed G5 (Gastrointestinal disorders) | 1 (1)
Cognitive disturbance G2 (Nervous system disorders) | 1 (1)
Acute pancreatitis G3 (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased G3 (Investigations) | 1 (1)
Alkaline phosphatase increased G3 (Investigations) | 1 (1)
AST incresed G3 (Investigations) | 1 (1)
ALT increased G3 (Investigations) | 1 (1)
GGT increased G3 (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib Arm (N=25)
Vomiting G1 (Gastrointestinal disorders) | 6 (6)
Intermittent vomiting G1 (Gastrointestinal disorders) | 4 (4)
Vomiting G2 (Gastrointestinal disorders) | 1 (1)
Vomiting G3 (Gastrointestinal disorders) | 1 (1)
Fatigue G1 (General disorders) | 5 (7)
Fatigue G2 (General disorders) | 8 (8)
Intermittent nausea G1 (Gastrointestinal disorders) | 3 (3)
Nausea G1 (Gastrointestinal disorders) | 6 (7)
Nausea G2 (Gastrointestinal disorders) | 1 (1)
Nausea G3 (Gastrointestinal disorders) | 1 (1)
Worsened back pain G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Jaw pain right G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Loss of consciousness, transient G1 (Nervous system disorders) | 1 (1)
Bilateral femur pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vaginal bleeding G1 (Reproductive system and breast disorders) | 1 (1)
Urinary tract infection G1 (Renal and urinary disorders) | 1 (1)
Shortness of breath G1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Worsened DOE G1 (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea G1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperkalemia G2 (Metabolism and nutrition disorders) | 1 (1)
Worsened anemia G1 (Blood and lymphatic system disorders) | 2 (2)
Worsened anemia G2 (Blood and lymphatic system disorders) | 1 (1)
Worsening anemia G3 (Blood and lymphatic system disorders) | 1 (1)
Anemia (secondary to GI bleed) G3 (Blood and lymphatic system disorders) | 1 (1)
Neutropenia G2 (Blood and lymphatic system disorders) | 2 (3)
Intermittent worsened abdominal pain w/ radiation to R shoulder G2 (Gastrointestinal disorders) | 1 (1)
Intermittent back pain G1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Worsened low back pain with radiation to buttocks, R hip G2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute lower back pain G2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent diarrhea G1 (Gastrointestinal disorders) | 2 (2)
Diarrhea G1 (Gastrointestinal disorders) | 9 (9)
Intermittent constipation G1 (Gastrointestinal disorders) | 2 (2)
Constipation G2 (Gastrointestinal disorders) | 1 (1)
Decreased appetite G1 (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite G2 (Metabolism and nutrition disorders) | 1 (1)
Anorexia G1 (Metabolism and nutrition disorders) | 2 (2)
Intermittent cramps abdomen G1 (Gastrointestinal disorders) | 1 (1)
Intermittent cramps, feet (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent pain/cramps legs G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain elbow G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Early satiety G1 (Gastrointestinal disorders) | 3 (3)
Intermittent night sweats G1 (General disorders) | 2 (2)
Hemorrhoids G1 (Gastrointestinal disorders) | 1 (1)
Facial flushing G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Generalized depigmentation G2 (Skin and subcutaneous tissue disorders) | 1 (1)
Decreased strength G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory symptoms G1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weakness lower extremities G2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized weakness G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight loss G1 (General disorders) | 2 (2)
Leukopenia G2 (Blood and lymphatic system disorders) | 1 (1)
Hypertension G1 (Vascular disorders) | 1 (1)
Hypertension G2 (Vascular disorders) | 6 (7)
Hypertension G3 (Vascular disorders) | 3 (4)
Epistaxis G1 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Constipation G1 (Gastrointestinal disorders) | 2 (2)
Pain B/L legs R>L G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased urine output (Renal and urinary disorders) | 1 (1)
Leukopenia G1 (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia G1 (Blood and lymphatic system disorders) | 1 (1)
Fever G1 (General disorders) | 1 (1)
Abdominal cramping G2 (Gastrointestinal disorders) | 1 (1)
Intermittent postprandial cramping G1 (Gastrointestinal disorders) | 1 (1)
Intermittent abdominal pain G1 (Gastrointestinal disorders) | 1 (1)
Abdominal pain G1 (Gastrointestinal disorders) | 4 (4)
Left lower abdominal and lower back pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain G2 (Gastrointestinal disorders) | 5 (6)
Pain G2 (General disorders) | 2 (2)
Worsened LUQ pain G3 (Gastrointestinal disorders) | 1 (1)
Axorexia G2 (Gastrointestinal disorders) | 1 (1)
Headache G1 (Nervous system disorders) | 6 (6)
Headache G3 (Nervous system disorders) | 1 (1)
Hand/foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Joint and muscle pain G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent right shoulder pain G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening pain G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Left wrist pain with cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower back and left calf pain G2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent leg cramps G1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Leg cramps (pain) G2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent sore mouth G1 (Gastrointestinal disorders) | 1 (1)
Mouth pain G1 (Gastrointestinal disorders) | 3 (3)
Oral dysesthesia G1 (Gastrointestinal disorders) | 1 (1)
Rhinorrhea and throat discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrush (mucosal infection) G1 (Infections and infestations) | 1 (1)
oral candidiasis G2 (Infections and infestations) | 1 (1)
Dysgeusia G1 (Gastrointestinal disorders) | 1 (1)
Hypomagnesemia G1 (Metabolism and nutrition disorders) | 3 (3)
Cystitis G1 (Renal and urinary disorders) | 1 (1)
Proteinuria G2 (Renal and urinary disorders) | 1 (1)
Proteinuria G3 (Renal and urinary disorders) | 1 (1)
Elevated UPC G1 (Renal and urinary disorders) | 1 (1)
Blood bilirubin increased G1 (Investigations) | 2 (2)
Blood bilirubin increased G2 (Investigations) | 1 (1)
Alkaline phosphatase increased G1 (Investigations) | 1 (1)
GGT increased G1 (Investigations) | 1 (1)
ALT increased G1 (Investigations) | 1 (1)
AST increased G1 (Investigations) | 2 (2)
AST increased G2 (Investigations) | 1 (1)
Alkaline phosphatase increased G2 (Investigations) | 1 (1)
GGT increased G2 (Investigations) | 1 (1)
Hypoalbuminemia G2 (Metabolism and nutrition disorders) | 1 (1)
Ascites G3 (Gastrointestinal disorders) | 1 (1)
Rash G1 (Skin and subcutaneous tissue disorders) | 3 (3)
Facial and hand edema G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Infection - rash G2 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation - perianal G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Hypopigmentation B/L forearms G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin dryness G1 (Skin and subcutaneous tissue disorders) | 2 (2)
Whitening of hair G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus G1 (Skin and subcutaneous tissue disorders) | 1 (1)
Hair lightening G2 (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety G1 (Psychiatric disorders) | 1 (1)
Insomnia G1 (Psychiatric disorders) | 1 (1)
Muscle weakness G1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Drowsiness G1 (General disorders) | 1 (1)
Cough G1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left ankle weakness G2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypothyroidism G2 (Endocrine disorders) | 1 (1)
Epistaxis G2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration G3 (General disorders) | 1 (1)
Retching G1 (Gastrointestinal disorders) | 1 (1)
Hypotension G3 (Vascular disorders) | 1 (1)
Lightheadedness G1 (General disorders) | 1 (1)
Dizziness G1 (General disorders) | 1 (1)
Bloating G1 (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes